CLINICAL TRIAL: NCT01350505
Title: Toileting at Night in Older Adults: Light to Maximize Vision, Minimize Insomnia
Brief Title: Toileting at Night in Older Adults: Light to Maximize Balance, Minimize Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: E0773-P
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Falls; Balance; Insomnia; Aging
Keywords: Postural Balance; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The order of the interventions were randomized to the four visits.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): 13 minutes of light at night (2 hours after bedtime)
  Interventions: Behavioral: White light exposure; Behavioral: Dim white light exposure; Behavioral: Very dim white light exposure; Behavioral: Dim orange light exposure

INTERVENTIONS:
Behavioral: White light exposure — ~200 lux of broad spectrum white light
Behavioral: Dim white light exposure — ~28 lux of broad spectrum white light
Behavioral: Very dim white light exposure — <0.5 lux of broad spectrum white light
Behavioral: Dim orange light exposure — ~28 lux of orange light

SUMMARY:
To examine the change in balance that occurs in older individuals when exposed to different colored lights at night.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-85
* Stable health
* Normal color vision

Exclusion Criteria:

* Alcohol abuse
* Depression
* Sleep disorders
* Smoking
* Use of illegal drugs

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Zeitzer, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All relevant summary data is presented in a publication under review. Anonymized, individual participant data would be made available upon request and completion of necessary documentation.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] McBean AL, Najjar RP, Schuchard RA, Hall CD, Wang CA, Ku B, Zeitzer JM. Standing Balance and Spatiotemporal Aspects of Gait Are Impaired Upon Nocturnal Awakening in Healthy Late Middle-Aged and Older Adults. J Clin Sleep Med. 2016 Nov 15;12(11):1477-1486. doi: 10.5664/jcsm.6270. PMID 27448415

RESULTS

PARTICIPANT FLOW:
Groups:
- Light Exposure: 13 minutes of experimental light exposure during the night
Period: Overall Study
Arm/Group | Light Exposure
Started | 21
Completed | 17
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Light Exposure
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 26.9 (6.1)
Baseline total sleep time [Mean (Standard Deviation); unit: hours] | 7.32 (.73)
Baseline sleep efficiency [Mean (Standard Deviation); unit: % of time in bed person is asleep] | 91.9 (5.6)
Balance Self-Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — 0-100, with higher scores being better balance
  units on a scale | 97.3 (3.0)
Mini Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — 0-30, with higher scores being better overall cognition
  units on a scale | 29.9 (0.3)
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — 0-21, with higher scores being worse sleep and scores >5 associated with clinically significant sleep problems
  units on a scale | 2.3 (1.4)
Geriatric Depression Scale [Mean (Standard Deviation); unit: units on a scale] — 0-15, with higher scores representing greater depressive symptoms; scores >5 are suggestive of depression and >10 are almost always depression
  units on a scale | 0.6 (0.9)
Alcohol Use Disorders Identification Test [Mean (Standard Deviation); unit: units on a scale] — 0-40, higher scores representing greater risk for alcohol use disorder
  score: 0-7, Alcohol education score 8-15, Simple advice score 16-19, Simple advice plus brief counseling and continued monitoring score 20-40, Referral to specialist for diagnostic evaluation and treatment
  units on a scale | 1.5 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Balance
Description: Balance was assessed during a 13-minute nocturnal light exposure (4 different conditions) and differences between the conditions were assessed. To determine goodness of balance while walking, the variability in stride length (i.e., variance in stride-to-stride length) was calculated in each of the conditions. Increased variability in stride length is associated with increased risk of falling.
Time Frame: 13 minutes
Population: Healthy older adults. Note 4 participants declined to participate in the last condition (white room light).
Measure: Mean (Standard Deviation); unit: %CV
Arm/Group | Light Exposure
Number analyzed (Participants) | 21
%CV
  Very Dim White - Step Length | 6.66 (3.08)
  Dim White - Step Length | 5.34 (2.00)
  Dim Orange - Step Length | 5.62 (2.52)
  Room White - Step Length: number analyzed (Participants) | 17
  Room White - Step Length | 5.78 (2.87)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 day
Description: The definition of "adverse" and "serious adverse events" that we used were the same as that on clinicaltrials.gov.
Arm/Group | Light Exposure
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
* Tested only at a single, approximate circadian phase
* Did not have a large enough sample size to discriminate the effect of awakening out of different sleep stages or the impact of factors such as age, sex, and race

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT01350505/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT01350505/SAP_001.pdf
  • Informed Consent Form (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT01350505/ICF_002.pdf